CLINICAL TRIAL: NCT01804686
Title: A Phase 3b, Multicenter, Open-label, PCI-32765 (Ibrutinib) Long-term Extension Study
Brief Title: A Long-term Extension Study of PCI-32765 (Ibrutinib)
Acronym: CAN3001
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Collaborators: Pharmacyclics LLC. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR100955; PCI-32765CAN3001 (Other: Janssen Research & Development, LLC); 2012-004225-24 (EudraCT Number)
Record Dates: First submitted 2013-03-04; First posted 2013-03-05 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma; Mantle Cell Lymphoma; Follicular Lymphoma; Diffuse Large B-cell Lymphoma; Waldenstrom Macroglobulinemia; Chronic Graft Versus Host Disease
Keywords: Chronic lymphocytic leukemia; Small lymphocytic lymphoma; Mantle cell lymphoma; Follicular lymphoma; Diffuse large B-cell lymphoma; PCI-32765; Ibrutinib; Bruton's tyrosine kinase inhibitor; IMBRUVICA; JNJ-54179060
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Mantle-Cell; Lymphoma, Follicular; Lymphoma, Large B-Cell, Diffuse; Waldenstrom Macroglobulinemia; Bronchiolitis Obliterans Syndrome | interventions — ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (1):
- Ibrutinib (Experimental)
  Interventions: Drug: Ibrutinib

INTERVENTIONS:
Drug: Ibrutinib — Ibrutinib will be given orally as capsules, once daily continuously, according to the current dosing regimen established in the parent ibrutinib clinical study (560 mg, 420 mg, 280 mg, or 140 mg), at approximately the same time each day.
  Other Names: PCI-32765

SUMMARY:
The purpose of this study is to collect long-term safety and efficacy data for participants treated with ibrutinib and to provide ongoing access to ibrutinib for participants who are currently enrolled in ibrutinib studies that have been completed according to the parent protocol, are actively receiving treatment with ibrutinib, and who continue to benefit from ibrutinib treatment.

DETAILED DESCRIPTION:
This is an open-label (identity of assigned study drug will be known) study designed to collect long-term safety and efficacy data and provide ibrutinib access to participants in completed ibrutinib studies. PCI-32765 (Ibrutinib) is a first-in-class, potent, orally-administered, covalently-binding small molecule inhibitor of bruton's tyrosine kinase. "PCI-32765" and "ibrutinib" refer to the same molecule; hereafter, "ibrutinib" will be used. Participants will continue with the current ibrutinib dosing regimen established in the parent ibrutinib study until the investigator determines that the participant is no longer benefitting from treatment (ie, disease progression or unacceptable toxicity has occurred), the participant withdraws consent, alternative access to ibrutinib is available and feasible (example, participant assistance program or commercial source of ibrutinib), or for other reasons as defined in the protocol, or until the end of the study, whichever occurs earlier. Safety will be monitored throughout the study and summarized. Efficacy may be analyzed in combination with the data collected in the parent protocol. There is no formal hypothesis testing planned for this long-term extension study. Participants for whom alternative access to ibrutinib is not available and feasible can receive treatment with single-agent ibrutinib until end of study, which is defined as the time when all participants still receiving study treatment have transitioned to commercial or alternative access to ibrutinib, have stopped receiving ibrutinib treatment, or upon a decision by the sponsor to terminate the study, whichever occurs earlier.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be currently participating in an ibrutinib clinical study considered complete and have received at least 6 months of treatment with ibrutinib. At study entry, participants must be actively receiving treatment with single-agent ibrutinib; or participants must have participated in an ibrutinib randomized clinical study in which they initially received comparator treatment and now cross-over to ibrutinib. Note: A minimum of 6 months requirement for prior ibrutinib treatment will not be mandatory in this case and participants with less than 6 months will be required to have more frequent initial safety assessments; or participants must be currently participating in study PCI-32765LYM1002. At study entry, participants must be actively receiving combination treatment with ibrutinib and nivolumab or single-agent ibrutinib
* Investigator's assessment that the benefit of continued ibrutinib therapy as a single agent or in combination with nivolumab will outweigh the risks
* Agrees to protocol-defined use of effective contraception
* Negative blood or urine pregnancy test at screening

Exclusion Criteria:

* Requires anticoagulation with warfarin or equivalent vitamin K antagonists
* Requires treatment with strong cytochrome P450 (CYP)3A4/5 inhibitors, unless previously approved by sponsor
* Any condition or situation which, in the opinion of the investigator, may put the participant at significant risk, may confound the study results, or may interfere significantly with volunteer's participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2013-09-09 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-01-29 (Estimated)

PRIMARY OUTCOMES:
Number of participants affected by an adverse event | Up to 30 days after the last dose of study drug, or until the start of a subsequent systemic anti-cancer therapy, if earlier

SECONDARY OUTCOMES:
Number of participants with change in disease status | Up to the end-of-treatment visit (up to 30 days after the last dose of study medication), or until the start of a subsequent anti-caner therapy, if earlier

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (174):
- United States (32):
  - City of Hope Cancer Center, Duarte, California
  - University of California San Diego Medical Center, La Jolla, California
  - University of California Los Angeles, Los Angeles, California
  - St. Joseph Hospital Center for Cancer Prevention and Treatment, Orange, California
  - Stanford University Medical Center, Stanford, California
  - Stanford University, Stanford, California
  - Norwalk Medical Group, Norwalk, Connecticut
  - Northwest Georgia Oncology Centers PC, Marietta, Georgia
  - Northwestern University Hospital, Chicago, Illinois
  - Indiana University, Goshen, Indiana
  - Kansas University Medical Center, Westwood, Kansas
  - Louisville Oncology Suburban - Norton Cancer Institute, Louisville, Kentucky
  - Dana Farber Cancer Center, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Battle Creek Health Systm, Battle Creek, Michigan
  - Karmanos Cancer Institute - Wayne State University, Detroit, Michigan
  - Washington University, St Louis, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Weill Medical College of Cornell University, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Southeastern Medical Oncology Center, Goldsboro, North Carolina
  - The Ohio State University- James Cancer Hospital, Columbus, Ohio
  - Willamette Valley Cancer Center, Eugene, Oregon
  - Kaiser Permanente, Portland, Oregon
  - University of Pennsylvania Medical Center, Philadelphia, Pennsylvania
  - Avera Medical Group, Sioux Falls, South Dakota
  - MD Anderson Cancer Center - University of Texas, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
  - University of Washington, Seattle, Washington
  - West Virginia University, Morgantown, West Virginia
  - University of Wisconsin Carbone Cancer Center - Wisconsin Institute for Medical Research, Madison, Wisconsin
- Argentina (2):
  - CEMIC Saavedra, Ciudad Autonoma Buenos Aires
  - Fundaleu, Ciudad de Buenos Aires
- Australia (8):
  - Royal Adelaide Hospital, Adelaide
  - John Fawkner Cancer Trial Centre, Coburg
  - Concord Hospital, Concord
  - Austin Health, Heidelberg
  - Peter MacCallum Cancer Institute, Melbourne
  - Royal Perth Hospital, Perth
  - Alfred Hospital, Prahran
  - Adventist Health Care Limited trading as San Clinical Trials Unit, Wahroonga
- Belgium (6):
  - UZA, Antwerp
  - A.Z. Sint Jan, Bruges
  - UCL - Saint Luc, Brussels
  - UZ Gent - departement oncologie, Ghent
  - UZ Leuven Gasthuisberg, Leuven
  - UCL Mont-Godinne, Yvoir
- Brazil (3):
  - Ministerio da Saude Instituto Nacional do Cancer, Rio de Janeiro
  - Santa Casa da Misericórdia da Bahia - Hospital Santa Isabel, Salvador
  - Instituto de Ensino e Pesquisa São Lucas, São Paulo
- Jewish General Hospital, Montreal, Quebec, Canada
- China (12):
  - Peking University People's Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - Peking University First Hospital, Beijing
  - West China Hospital Sichuan University, Chengdu
  - Fujian Medical University, Fuzhou
  - Sun Yat-sen University Cancer Hospital, Guangzhou
  - Zhejiang University First Hospital, Hangzhou
  - Ruijin Hospital, Shanghai
  - Tangdu hospital the Fourth Military Medical, Shanxi
  - The First Affliated Hospital of Soochow University, Suzhou
  - The Institute of Hematological disease, Tianjin
  - Wuhan Union Hospital, Wuhan
- Colombia (2):
  - Fundacion Santa Fe, Bogotá
  - Fundacion Oftalmologica de Santander - FOSCAL, Floridablanca
- Czechia (3):
  - Fakultni nemocnice Brno, Interni hematologicka a onkologicka klinika, Brno
  - Fakultni nemocnice Kralovske Vinohrady - Interni hematologicka klinika, Prague
  - Vseobecna fakultni nemocnice v Praze - I. interni klinika - klinika hematologie, Prague
- France (7):
  - Hopital Henri Mondor, Créteil
  - Hôpital E. Muller, Mulhouse
  - HOPITAL SAINT LOUIS - Hematology / Oncology, Paris
  - Hopital Necker Enfants Malades, Paris
  - Hopital Haut Leveque Service Maladie Du Sang, Pessac
  - CH LYON SUD - Hematology, Pierre-Bénite
  - CHU de Tours, Tours
- Germany (9):
  - Vivantes Klinikum Spandau-Klinik f. Innere Medizin Hämatologie/Onkologie/Gastroenterologie - Germany, Berlin
  - Universitätsklinikum Carl Gustav Carus; Med. Klinik und Poliklinik I - Hämatologische Ambulanz, Haus, Dresden
  - Universitätsklinikum Essen; Klinik f. Hämatologie- Germany, Essen
  - Justus-Liebig-Universitaet - Medizinische Klinik IV, Haematologie, Giessen
  - Universitätsklinikum Heidelberg Med. Klinik IV, Heidelberg
  - Universitätsklinikum des Saarlandes, Homburg/Saar
  - Gemeinschaftspraxis Dres. Uhle/Müller/Kröning/Jentsch-Ullrich - Germany, Magdeburg
  - OnkoNet Marburg GmbH, Marburg
  - Universitätsklinikum für Innere Med. III_Hämatologie, Onkologie...- Germany, Ulm
- Greece (2):
  - Laiko General Hospital - 1st department of Internal Medicine, Athens
  - G Papanikolaou Hospital of Thessaloniki, Thessalonikis
- Hungary (2):
  - Semmelweis Egyetem, I. Belgyogyaszati Klinika, Budapest
  - Szegedi Tudomanyegyetem II. Belgyogyaszati Klinika, Szeged
- St James's Hospital, Dublin, Ireland
- Israel (6):
  - Haemek Medical Center, Afula
  - Hillel Yaffe Medical Center - Oncology, Hadera
  - Rambam Health Care Campus, Haifa
  - Rabin Medical Center Beilinson Campus, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (3):
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - DIPARTIMENTO DI BIOTECNOLOGIE CELLULARI ED EMATOLOGIA - UNIVERSITà ''LA SAPIENZA'', Roma
  - A.O.Citta della Salute e della Scienza di Torino, Torino
- Japan (3):
  - Tokyo Metropolitan Cancer and Infectious Diseases Center Komagome Hospital, Bunkyō City
  - Hiroshima University Hospital, Hiroshima
  - Hokkaido University Hospital, Sapporo
- Oaxaca Site Management Organization S.C., Oaxaca City, Mexico
- VU medisch centrum - Afd.Interne - INT, Amsterdam, Netherlands
- Poland (7):
  - Szpital Specjalistyczny w Brzozowie Podkarpacki Osrodek Onkologiczny im Ks B Markiewicza, Brzozów
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej Zespol Szpitali Miejskich, Chorzów
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Pratia MCM Krakow, Krakow
  - Oddzial Hematologii, Opole
  - Wojewodzki Szpital Specjalistyczny im. Janusza Korczaka, Słupsk
  - Katedra I Klinika Hematologii Nowotworow Krwi I Transplantacji Szpiku, Wroclaw
- Portugal (3):
  - Instituto Portugues de Oncologia, Lisbon
  - Hospital De Santa Maria, Lisbon
  - Instituto Portugues de Oncologia, Porto
- Auxilio Mutuo Cancer Center, San Juan, Puerto Rico
- Russia (18):
  - Arkhangelsk Regional Clinical Hospital, Arkhangelsk
  - Chelyabinsk Regiona Onc. Center, Chelyabinsk
  - Emergency Hospital of Dzerzhinsk, Dzerzhinsk
  - Cancer Research Center, Moscow
  - S.P. Botkin Moscow City Clinical Hospital, Moscow
  - Regional Clinical Hospital n.a.Semashko, Nizhny Novgorod
  - Medical Scientific Radiology - Center, Obninsk
  - Perm Medical Sanitary Unit#1, Perm
  - Republican Hospital named by V.A.Baranova, Petrozavodsk
  - Rostov Research Institute of Oncology, Rostov-on-Don
  - Ryazan Regional Clinical Hospital, Ryazan
  - Clinical Research Institute of Hematology and Transfusiology, Saint Petersburg
  - Federal Center of Heart, Blood and Endocrinology, Saint Petersburg
  - City Clinical Oncology Dispensary, Saint Petersburg
  - Leningrad region clinical hospital, Saint
  - Samara Region Clinical Hospital, Samara
  - Oncological dispensary #2, Sochi
  - Oncology Dispensary of Komi Republic, Syktyvkar
- South Korea (2):
  - National Cancer Center, Goyang-si
  - The Catholic University of Korea Seoul St Mary s Hospital, Seoul
- Spain (8):
  - Hospital Vall d'Hebron, Barcelona
  - Inst. Cat. Doncologia-H Duran I Reynals, L'Hospitalet de Llobregat
  - Hosp. Univ. de La Princesa, Madrid
  - Hosp. Gral. Univ. Gregorio Maranon, Madrid
  - Hosp. Univ. Infanta Leonor, Madrid
  - Fundacion Jimenez Diaz, Madrid
  - Clinica Universitaria de Navarra, Pamplona
  - Hospital Clinico Universitario Salamanca, Salamanca
- Sweden (3):
  - Sahlgrenska University hospital, Hematology Dept, Gothenburg
  - Skanes universitetssjukhus, Lund
  - Karolinska Universitetssjukhuset Solna, Centrum för Hematologi, Stockholm, Stockholm
- Changhua Cristian Hospital, Changhua County, Taiwan
- Turkey (Türkiye) (5):
  - Ankara University, Ankara
  - American Hospital, Istanbul
  - Istanbul University, Istanbul
  - Dokuz Eylul Universitesi Tip Fakultesi, Izmir
  - Erciyes University, Kayseri
- Ukraine (7):
  - Communal Nonprofit Enterprise 'Cherkasy Regional Oncology Dispensary Of Cherkasy Regional Council', Cherkasy
  - Dnepropetrovsk City Clinical Hospital #4, Regional Hematology Center, Dnipro
  - SI Grigoriev Institute for Medical Radiology National Academy of Medical Science of Ukraine, Kharkiv
  - Khmelnitskiy Regional Hospital, Hematology Department, Khmelnitskiy
  - State Institution Scientific Center for Radiation Medicine Academy of Medical Sciences of Ukraine, Kiev
  - Institute of Blood Pathology and Transfusion Medicine of AMS of Ukraine, Lviv
  - Vinnytsya Regional Clinical Hospital named after M.I.Pirogov, Vinnitsa
- United Kingdom (15):
  - University Hospitals Birmingham NHS Trust,, Birmingham
  - Royal Bournemouth Hospital, Bournemouth
  - Colchester Hospital University NHS, Colchester
  - Beatson West Of Scotland Cancer Centre, Glasgow
  - St James's Institute of Oncology, Leeds
  - Leicester Royal Infirmary - Haematology, Leicester
  - St Bartholomew's Hospital - Dept of Haematology, London
  - University College London Hospitals NHSFT, London
  - Kings College Hospital, London
  - Christie Hospital, Manchester
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Derriford Hospital, Plymouth
  - Royal Hallamshire Hospital, Sheffield
  - Southampton General Hospital, Southampton
  - Royal Marsden Hospital (Sutton), Sutton